CLINICAL TRIAL: NCT04899726
Title: Description of the Safety and Functionality of a Rectoscope (P201630551) That Allows the Identification of the Distal Section Margin in Oncological Rectal Surgery
Brief Title: Description of the Safety and Functionality of a Rectoscope (P201630551)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P201630551
Record Dates: First submitted 2021-05-21; First posted 2021-05-24 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Oncological Rectal Surgery
MeSH Terms: interventions — Proctoscopes

STUDY DESIGN:
Intervention Model Description: Pilot Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Oncology patients candidate for rectal surgery (tumors located up to 15 cm from the anal margin) and meet inclusion criteria. Rectoscope (P201630551) allows the identification of the distal section margin.
  Interventions: Device: Rectoscope (P201630551)

INTERVENTIONS:
Device: Rectoscope (P201630551) — Rectoscope (P201630551) allows the identification of the distal section margin in oncological rectal surgery.

SUMMARY:
Most patients with rectal cancer receive neoadjuvant therapy. This usually causes a decrease in tumor size. In approximately 20% of patients who receive neoadjuvant therapy, the tumor disappears completely (complete pathological response), showing as a scar on the rectal mucosa, not noticeable from the rectal serosa, from outside the rectum, difficulting the identification of the tumor location by the surgeon.

Rectoscope (p201630551) allows the surgeon to view the illuminated rectum from the patient's abdomen, determining the appropriate point of section of the rectum.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18 years old.
* Patients with rectal cancer (15 cm or less from the anal margin), whether or not they have received neoadjuvant treatment, in whom cancer surgery is to be performed through the anterior (abdominal) route, whether laparoscopic or not.
* Patients who accept their participation in this study, after explaining the study details.
* Patients who sign the informed consent.

Exclusion Criteria:

* Patients who are going to undergo an abdominoperineal amputation or transanal surgery for rectal cancer.
* Patients who do not accept their participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-07-14 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events related to use of the device. | at immediate postoperative period
  Safety. Clavien-Dindo classification will be used.
Evaluation of functionality | at surgery
  Categorical variable. 3 options:
  1. the device has worked without problems
  2. the device has worked, but with problems
  3. the device could not carry out its function.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario La Paz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No